CLINICAL TRIAL: NCT05006976
Title: A Naturalistic Trial of Nudging Patients and Clinicians in the Norwegian Sickness Absence Clinics- The NSAC Nudge Study
Brief Title: A Naturalistic Trial of Nudging Clinicians in the Norwegian Sickness Absence Clinic. The NSAC Nudge Study
Acronym: NSAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University Hospital of North Norway (Other); Opptreningssenteret i Finnmark (Alta, Norway) (Unknown); Helgeland Hospital Trust (Other); Finnmarkssykehuset HF (Kirkenes, Norway) (Unknown); UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSAC Nudge
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-08

CONDITIONS: Musculoskeletal Disorder; Anxiety Disorders; Depression; Fatigue; Pain; Occupational Exposure; Work Related Stress; Workplace Bullying; Employment; Sickness Absence; Return to Work
Keywords: Return to work; Sickness absence; Nudge; Barriers for return to work; Motivation for work; Demand and control; Work/family conflict; Bullying
MeSH Terms: conditions — Musculoskeletal Diseases; Anxiety Disorders; Depression; Fatigue; Pain; Occupational Stress; Bullying

STUDY DESIGN:
Intervention Model Description: Patients are randomized in equal proportions to fill out either of two different questionnaires, consisting either of 1) health related questions only or 2) health related questions as well as questions concerning motivation for work, barriers for return to work and work environment. In both treatment arms, clinicians receive a summary of patient survey information on mental health and musculoskeletal pain. In the intervention arm, clinicians are nudged to have particular attention towards motivation for work, barriers for return to work and work environment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant is masked to which questionnaire he/she fills out. The primary outcome is functional recovery, operationalized in the short term as prevention of sickness absence or return to work, and in the long term as employment or disability benefits. To this end, registry data on employment status or qualification for disability benefits is applied. Clinicians (usually the patient's general practitioner) and case managers involved in decisions on medically certified sickness absence and disability benefits are blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSAC health only (Active Comparator): Treatment as usual (TAU) at NSAC, following a digital survey of health problems and the provision of a condensed report of this survey to clinician prior to consultation.
  Interventions: Other: NSAC health only
- NSAC health + MBW (Experimental): Treatment as usual (TAU) at NSAC, following a digital survey of health problems as well as Motivation, Barriers for return to work and Work environment (MBW), and the provision of a condensed report of this survey to clinician prior to consultation.
  Interventions: Other: NSAC health + MBW

INTERVENTIONS:
Other: NSAC health only — NSAC is an outpatient service delivered under the auspices of the specialist health care sector to patients currently on sick leave or at risk for long-term sickness absence. The service is staffed by medical doctors specialising in musculoskeletal health, physiotherapists, psychologists and welfare sector counsellors, and aims to provide patients with multi-disciplinary treatment with the intent of functional recovery. In "NSAC health only", clinicians are provided survey information on potential health problems only.
  Arms: NSAC health only
Other: NSAC health + MBW — NSAC is an outpatient service delivered under the auspices of the specialist health care sector to patients currently on sick leave or at risk for long-term sickness absence. The service is staffed by medical doctors specialising in musculoskeletal health, physiotherapists, psychologists and welfare sector counsellors, and aims to provide patients with multi-disciplinary treatment with the intent of functional recovery. In "NSAC health + MBW" clinicians are provided survey information on potential health problems as well as information on motivation for work, barriers for return to work and work environment factors.
  Arms: NSAC health + MBW

SUMMARY:
The Norwegian Sickness Absence Clinic (NSAC) Nudge Study is a naturalistic randomized controlled multicentre trial which aim is to measure the efficacy of nudging clinicians' attention towards patients' motivation for work, barriers for return to work and work environment challenges, on functional recovery as primary outcome, and health outcomes as secondary outcome.

Patients will be recruited in five different NSACs across northern Norway. In total 1100 patients will be randomized to two equal probability treatment arms: 1) NSAC with the nudge, and 2) NSAC without the nudge. The nudge is tailored to the individual patient's needs using survey, and the clinicians are presented with a summary of this patient survey prior to consultations highlighting health problems and challenges as reported by the patient in the survey.

DETAILED DESCRIPTION:
The NSAC Nudge Study is part of a broader project, the Norwegian Sickness Absence Clinic Study (NSACS). The NSACS has two sources of funding (Northern Norway Regional Health Authority and The Norwegian Labour and Welfare Administration (NAV)), and involves two RCTs (NSAC Nudge and NSAC Efficacy) and fifteen work packages covering aspects of efficacy, interactions in efficacy, scalability, health economics, and characteristics of the target group and the patient group. The randomized controlled trial (RCT) NSAC Nudge is the subject of this trial registration. A list of the associated work-packages (WPs) is available in the protocol attached this registration at a later time point.

The NSAC Nudge Study is a randomized controlled multicentre trial, carried out in northern Norway and involving 5 Norwegian Sickness Absence Clinics (NSAC [Helse i Arbeid]). The study will recruit 1100 patients, randomized in equal proportions to either of two treatment arms 1) Treatment at the NSAC following a patient survey of health problems and 2) treatment at the NSAC following a patient survey of health problems as well as a survey on motivation for work, barriers for return to work and work environment (MBW).

The NSACs are staffed by teams of medical doctors specializing in physical medicine and rehabilitation, psychologists, physiotherapists and employment support supervisors. The NSAC service aims to provide quick clarification of health problems or treatment to patients with common mental disorders or musculoskeletal health problems with the goals of functional improvement, prevention of long-term sickness absence and return to work.

All patients are asked to fill out an online survey about their health and MBW factors between time of referral and their first treatment. The survey will also handle randomization. The NSAC clinicians are given a summary to be used in the treatment of the individual patient, and the effect of this comprehensive mapping and the provision of a condensed report to clinician prior to consultation is the primary aim of the RCT. The clinicians will be trained in how providing this information is going to guide clinical practice and using this information in treatment of patients.

The anticipated mechanism of the nudge is 1) an increased expectation among patients that MBW factors will be addressed during treatment, and/or 2) an increased focus on MBW factors by clinician in treatment, both due to the report and the patients' expectations. Whether this mechanism has an effect on patients' return to work (RTW) outcomes, prevention of sickness absence and general alleviation of symptoms will also be explored.

The data necessary to answer the research questions are gathered from national registries via personal identifier, registry data on population level, questionnaires filled out by the patient (data on health and working conditions) and questionnaires filled out by the clinician after each consultation (data on number of treatments, diagnosis, professions involved and types of treatment provided).

The patient questionnaire is divided in two surveys; 1) a health survey and 2) a survey on health and MBW. The health survey covers health, and includes musculoskeletal problems, mental health and other health related issues (such as alcohol consumption, medication and physical activity). The MBW survey includes working conditions (including inter alia questions on social support, work/family conflict and bullying), barriers for RTW, labour market affiliation, other personal aspects (such as demography and motivation for work), questionnaires for health economic evaluation and expectations for treatment.

By and large the questionnaire consists of test batteries which have been validated for specific topics. In an effort to reduce the number of questions posed to each patient, the baseline questionnaire will employ index questions which have proven psychometric properties in terms of factor loading or similar, meaning that if a problem on a specific topic such as neck pain is not indicated, the patient will not be presented with the Neck Disability Index questionnaire. The patient questionnaires will be filled out electronically after referral and prior to first treatment (Baseline, Time 0), as well as at 6 months after baseline (Time 1). We planned for a 12-month follow-up survey, but because of a technical error this second survey was never sent to participants. Accordingly the second follow-up survey will be sent to participants ultimo June 2024, which is in the interval between 17- and 31 months (depending on date of recruitment) after time of baseline survey (Time 2).

In the NSAC Nudge Study, receiving treatment at NSAC (Norwegian name HiA) does not presuppose consent to participate in research, but a mapping of health status is nevertheless a mandatory part of treatment. However, participation in research requires sharing these data and access to registry-based data for the involved patients.

ELIGIBILITY:
Inclusion Criteria:

* For the study, the single inclusion criteria is that the patient is offered a consultation or treatment at the NSAC (Norwegian: HiA).

Exclusion Criteria:

* Aged younger than 23 years at time of referral. The NSACs have guidelines that describe eligibility for treatment, and excludes patients that are either too healthy for the measure, too sick for the measure, not relevant diagnosis or otherwise not considered being in the target group for the measure.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2028-04-12 (Estimated); Study Completion 2033-01-12 (Estimated)

PRIMARY OUTCOMES:
Functional recovery: status, plan and prognosis for employment versus sickness absence | At last appointment at NSAC (can vary substantially between patients, but generally < 3 months after first appointment at NSAC)
  Clinician report at last consultation of current status, plan and prognosis for patient employment versus sickness absence. Status is current employment versus sickness absence, plan refers to patients own ambition and plans for employment versus sickness absence short term, while prognosis refers to the clinicians assessment of prognosis for employment versus sickness absence in 12 months.
Functional recovery: sickness absence self-report | Up to 31 months post baseline survey
  Employment, sickness absence and application for rehabilitation benefits between Time 0 and Time 2, based on patient self-report.
Functional recovery: sickness absence registry data | 12 months post baseline survey
  Employment, sickness absence and application for rehabilitation benefits during first 365 days post baseline survey, based on registry data.
Functional recovery: disability benefits | 60 months post baseline survey
  Employment, sickness absence, rehabilitation benefits and disability benefits during 5-year period post baseline survey, all based on registry data.

SECONDARY OUTCOMES:
Mental health | Up to 31 months post baseline survey
  Changes in self-reported mental health between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Hopkins Symptoms Checklist - 10 (HSCL-10).
Anxiety | Up to 31 months post baseline survey
  Changes in self-reported anxiety between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Beck Anxiety Inventory (BAI). The instrument is provided to patients upon indication, defined as a HSCL-10 score > 1.4
Depressive symptoms | Up to 31 months post baseline survey
  Changes in self-reported depression between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Beck Depression Inventory (BDI). The instrument is provided to patients upon indication, defined as a HSCL-10 score > 1.4
Sleep | Up to 31 months post baseline survey
  Changes in self-reported sleep between Time 0 and Time 1, and between Time 0 and Time 2, measured using 3 questions commonly used to diagnose sleeping disorder according to the DSM-IV criteria for insomnia.
Health Anxiety | Up to 31 months post baseline survey
  Changes in self-reported health anxiety between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Whitely Index. All patients are asked the first question in the test battery, and the entire instrument is provided to patients with a score of >3 on this question
Subjective health complaints | Up to 31 months post baseline survey
  Changes in subjective health between Time 0 and Time 1, and between Time 0 and Time 2, measured using a modified version of the Ursin Health Inventory.
Back pain | Up to 31 months post baseline survey
  Changes in self-reported back pain Time 0 and Time 1, and between Time 0 and Time 2, measured using the Oswestry Disability Index (ODI). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain. In case of back pain, patients are provided the ODI.
Neck pain | Up to 31 months post baseline survey
  Changes in self-reported neck pain between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Neck Disability Index (NDI). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain. In case of neck pain, patients are provided the NDI.
Pain intensity | Up to 31 months post baseline survey
  Changes in self-reported pain intensity between Time 0 and Time 1, and between Time 0 and Time 2, measured using a visual analogue scale scored between 0 and 10. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on pain intensity during rest and activity.
Fear avoidance | Up to 31 months post baseline survey
  Changes in self-reported fear avoidance between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Fear Avoidance Beliefs Questionnaire (FABQ). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided the FABQ.
Physical activity | Up to 31 months post baseline survey
  Changes in self-reported level of physical between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Saltin-Grimby Physical Activity Level Scale (SGPALS).
Fatigue | Up to 31 months post baseline survey
  Changes in self-reported fatigue between Time 0 and Time 1, and between Time 0 and Time 2, measured using the Fatigue Assessment Scale. All patients are asked the first question in the test battery, and the entire instrument is provided to patients with a score of ≥ 3 on this question
Pain localization | Up to 31 months post baseline survey
  Changes in self-reported localization of pain between Time 0 and Time 1, and between Time 0 and Time 2. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain.
Cause of pain | Up to 31 months post baseline survey
  Changes in self-reported cause of pain between Time 0 and Time 1, and between Time 0 and Time 2. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on the believed cause of pain.
Self-reported diagnoses | Up to 31 months post baseline survey
  Changes in self-reported diagnoses between Time 0 and Time 1, and between Time 0 and Time 2. The respondent is asked whether he/she thinks they have Covid-19 sequelae, myalgic encephalomyelitis/chronic fatigue syndrome, whiplash, fibromyalgia, hypermobility, irritable bowel syndrome or food intolerance, or whether they have been diagnosed with either of these by health personnel.

OTHER OUTCOMES:
Preventive effect of sickness absence | Up to 31 months post baseline survey
  Changes in self-reported beliefs about the potential preventive effect of short-term sickness absence on long term sickness absence between Time 0 and Time 1, and between Time 0 and Time 2. The respondent is asked whether he/she agrees to 5 different statements on this topic, using a 5-point likert scale.
Health economic evaluation: self report | Up to 31 months post baseline survey
  Health economic evaluation is measured using the EQ-5D and the ReQol instruments, issued to patients at baseline (Time 0) and at Time 1 and Time 2, to assess change.
Health economic evaluation: labour costs | 12 months post baseline survey
  Health economic evaluation also involves data on number of professions seeing the patient and number of working hours spent on the patient by each profession seeing the patient during the treatment period, recorded in questionnaires filled out by the clinicians after each consultation. This enables calculation of costs in terms of manpower and staff.
Expectations to- and evaluation of treatment | Up to 31 months post baseline survey
  Using open-ended questions, patients are asked about their expectations towards treatment prior to first treatment, and about their evaluation of treatment 6- and 12 months first treatment. These two will be compared.
Barriers for return to work | Up to 31 months post baseline survey
  Changes in self-reported barriers for return to work between Time 0 and Time 1, and between Time 0 and Time 2. The questionnaire includes 26 items concerning barriers for return to work and is part of the survey in the MBW intervention.
Motivation for work | Up to 31 months post baseline survey
  Changes in self-reported motivation for work between Time 0 and Time 1, and between Time 0 and Time 2. The questionnaire consists of a number of questions concerning motivation, and is part of the survey in the MBW intervention.
Effort/reward imbalance | Up to 31 months post baseline survey
  Changes in self-reported effort/reward imbalance between Time 0 and Time 1, and between Time 0 and Time 2. Effort/reward imbalance is part of the survey in the MBW intervention, and is measured using the 3 items with the highest factor loading in the Siegrist Effort/Reward Imbalance Questionnaire (short version). A high score on either of the three items triggers the rest of the questionnaire.
Workplace bullying | Up to 31 months post baseline survey
  Changes in self-reported workplace bullying between Time 0 and Time 1, and between Time 0 and Time 2. Workplace bullying is measured using the Short Negative Acts Questionnaire (SNAQ).
Economic situation | Up to 31 months post baseline survey
  Changes in self-reported economic situation between Time 0 and Time 1, and between Time 0 and Time 2. The questionnaire includes 2 items concerning economic problems and concerns about economic problems.
Procedural justice | Up to 31 months post baseline survey
  Changes in self-reported procedural justice between Time 0 and Time 1, and between Time 0 and Time 2. Procedural justice is part of the survey in the MBW intervention, and is measured by 3 items concerning workplace decisions.
Relational justice | Up to 31 months post baseline survey
  Changes in self-reported relational justice between Time 0 and Time 1, and between Time 0 and Time 2. Relational justice is part of the survey in the MBW intervention, and is measured by 4 items concerning the general behaviour of the respondent's supervisor.
Job phobia | Up to 31 months post baseline survey
  Changes in self-reported job phobias between Time 0 and Time 1, and between Time 0 and Time 2. Job phobia is measured by 12 items concerning the respondent's avoidance of the workplace or work-related anxiety.
Ergonomic work environment | Up to 31 months post baseline survey
  Changes in self-reported ergonomic work environment between Time 0 and Time 1, and between Time 0 and Time 2. Ergonomic work environment is measured by 11 items concerning the respondent's physical tasks at work.
Organisational change | Up to 31 months post baseline survey
  Changes in self-reported organisational change between Time 0 and Time 1, and between Time 0 and Time 2. Organisational change is part of the survey in the MBW intervention, and is measured using the 3 items covering changes in management, colleagues and tasks.
Work/family conflict | Up to 31 months post baseline survey
  Changes in self-reported work/family conflict between Time 0 and Time 1, and between Time 0 and Time 2. Work/family conflict is part of the survey in the MBW intervention, and is measured using the 4 items with the highest factor loading in the Home-Work Interference Scale.
Demand and control | Up to 31 months post baseline survey
  Changes in self-reported demand and control between Time 0 and Time 1, and between Time 0 and Time 2. Demand and control is measured using three questions from the instrument developed by Karasek/Theorell, and is part of the survey in the MBW intervention. A high score on either of the three items triggers the rest of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arnstein Mykletun, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (5):
- Norway (5):
  - Helse I Arbeid Nordlandssykehuset, Bodø, Nordland
  - Helse I Arbeid Helgelandssykehuset, Sandnessjøen, Nordland
  - Opptreningssenteret i Finnmark, Alta, Troms Og Finnmark
  - Helse I Arbeid Finnmarkssykehuset, Kirkenes, Troms Og Finnmark
  - Helse I Arbeid Universitetssykehuset Nord-Norge, Tromsø, Troms Og Finnmark

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data with other researchers. At the stage of analyses, associated researchers will be provided with an anonymized data set including all relevant data to answer the research questions.

REFERENCES:
- [Derived] Bardal I, Aars NAP, Trichet LO, Brandseth OL, Terjesen C, Irgens E, Hansen BO, Kristoffersen A, Hoper A, Jenssen OR, Brinchmann B, Mykletun A. Expanding the Focus on Work Factors in an Outpatient Setting: Does a Nudge of Patients and Clinicians have an Effect on Return-to-Work and Benefits? Findings from the NSAC Nudge Multicentre Randomised Controlled Trial. J Occup Rehabil. 2025 Dec 12. doi: 10.1007/s10926-025-10343-x. Online ahead of print. PMID 41385138
- [Derived] Aars NA, Bardal I, Brinchmann B, Mykletun A. Naturalistic trial of nudging patients and clinicians in the Norwegian sickness absence clinics: a study protocol for the NSAC Nudge Study. BMJ Open. 2025 Mar 3;15(3):e089758. doi: 10.1136/bmjopen-2024-089758. PMID 40032398